CLINICAL TRIAL: NCT04675515
Title: CORE: CO Monitoring for Reach and Efficacy in Tobacco Treatment for Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Joseph D. Phillips, MD., Staff Physician, Thoracic Surgery, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D21008
Record Dates: First submitted 2020-12-11; First posted 2020-12-19 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2024-09

CONDITIONS: Tobacco Use; Cancer
MeSH Terms: conditions — Tobacco Use; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Tobacco Treatment (No Intervention): All individuals who are identified as tobacco users are offered tobacco treatment which includes proactive, as needed, contacts via in person, telehealth or telephone visits. for tobacco treatment, pharmacotherapy as indicated, and Quitline and SmokefreeTXT referrals
- Intensive Tobacco Treatment (Experimental): Patients who consent to study participation will meet with a tobacco treatment specialist in-person initially, then biweekly via telephone or telehealth or face-to-face (or more frequently as needed). They will receive tobacco treatment counseling and support from certified tobacco treatment specialist, which may include pharmacotherapy as indicated. At enrollment, participants will undergo carbon monoxide testing using a carbon monoxide monitor. At baseline, participants will complete the Fagerström Test for Nicotine Dependence, and the Cancer Patient Tobacco Use Questionnaire (C-TUQ).
  These tobacco related survey measures will be completed at 3 additional time points: 30 days, 3 months and 6 months.
  Interventions: Behavioral: Intensive Tobacco Treatment

INTERVENTIONS:
Behavioral: Intensive Tobacco Treatment — Bi-weekly tobacco treatment counseling and regular carbon monoxide monitoring
  Arms: Intensive Tobacco Treatment

SUMMARY:
The purpose of this study is to assess the cessation success rates of an intensive tobacco treatment program in a patients undergoing cancer treatment at 30 days, 3 months and 6 months.

DETAILED DESCRIPTION:
This mixed-methods, observational cohort study will assess intensive tobacco treatment with carbon monoxide monitoring offered to all eligible smoking patients presenting for cancer treatment to the NCCC at our main Lebanon campus and our very rural St. Johnsbury campus. Subjects will not be randomized and study will not be blinded. Cessation rates among the intensive tobacco treatment will be compared to usual care, matched historical controls, and to patients who refuse all tobacco treatment program elements.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and older
* Active Smoker at the time of initial consultation for cancer (defined as any smoking within 2 weeks of consult)

Exclusion Criteria:

* Adults unable to consent
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Change is smoking status | 30 days, 3 Months, 6 Months
  Change in smoking status (from smoking to not smoking) of those in an intensive tobacco treatment program at 30 days, 3 months and 6 months

SECONDARY OUTCOMES:
Motivational Impact of real-time carbon monoxide monitoring | 6 Months
  Motivational impact of real-time carbon monoxide monitoring in patients receiving intensive tobacco treatment as determined by a Motivation to Quit Assessment Questionnaire
Engagement Level with Tobacco Treatment via Telehealth | 6 Months
  Level of engagement with tobacco treatment via telehealth compared to historical control face-to-face visits as determined by a Technology Access and Experiences Questionnaire

OTHER OUTCOMES:
Engagement Level With Tobacco Treatment for Low Resource Patients outh! | 6 Months
  Level of engagement with tobacco treatment for low-resource patients who are provided cell phones with data plans as determined by a Technology Access and Experiences Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Phillips, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuan C, Morales-Oyarvide V, Babic A, Clish CB, Kraft P, Bao Y, Qian ZR, Rubinson DA, Ng K, Giovannucci EL, Ogino S, Stampfer MJ, Gaziano JM, Sesso HD, Cochrane BB, Manson JE, Fuchs CS, Wolpin BM. Cigarette Smoking and Pancreatic Cancer Survival. J Clin Oncol. 2017 Jun 1;35(16):1822-1828. doi: 10.1200/JCO.2016.71.2026. Epub 2017 Mar 30. PMID 28358654
- [Background] Duan W, Li S, Meng X, Sun Y, Jia C. Smoking and survival of breast cancer patients: A meta-analysis of cohort studies. Breast. 2017 Jun;33:117-124. doi: 10.1016/j.breast.2017.03.012. Epub 2017 Mar 31. PMID 28371644
- [Background] Sharp L, McDevitt J, Brown C, Carsin AE, Comber H. Association between smoking at diagnosis and cause-specific survival in patients with rectal cancer: Results from a population-based analysis of 10,794 cases. Cancer. 2017 Jul 1;123(13):2543-2550. doi: 10.1002/cncr.30583. Epub 2017 Mar 15. PMID 28297071
- [Background] Tammemagi CM, Neslund-Dudas C, Simoff M, Kvale P. Smoking and lung cancer survival: the role of comorbidity and treatment. Chest. 2004 Jan;125(1):27-37. doi: 10.1378/chest.125.1.27. PMID 14718417
- [Background] Fay KA, Phillips JD, Hasson RM, Fannin A, Millington TM, Finley DJ. Outcomes of an Intensive, Preoperative Smoking Cessation Program. Ann Thorac Surg. 2020 Feb;109(2):e137-e139. doi: 10.1016/j.athoracsur.2019.08.075. Epub 2019 Oct 3. PMID 31586615
- [Background] Phillips JD, Fay KA, Ramkumar N, Hasson RM, Fannin AV, Millington TM, Finley DJ. Long-Term Outcomes of a Preoperative Lung Resection Smoking Cessation Program. J Surg Res. 2020 Oct;254:110-117. doi: 10.1016/j.jss.2020.04.005. Epub 2020 May 16. PMID 32428728
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Land SR, Warren GW, Crafts JL, Hatsukami DK, Ostroff JS, Willis GB, Chollette VY, Mitchell SA, Folz JN, Gulley JL, Szabo E, Brandon TH, Duffy SA, Toll BA. Cognitive testing of tobacco use items for administration to patients with cancer and cancer survivors in clinical research. Cancer. 2016 Jun 1;122(11):1728-34. doi: 10.1002/cncr.29964. Epub 2016 Mar 28. PMID 27019325
- See also: Covita. Smokerlyzer. 2020 — https://www.covita.net/the-smokerlyzer-range/